CLINICAL TRIAL: NCT07337135
Title: Opioid-free Anesthesia vs Opioid-based Anesthesia / A Heavyweight Showdown - Randomized Controlled Trial
Brief Title: Opioid-Free vs Opioid-Based Anesthesia in Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital dos Lusíadas (Other)
Responsible Party: Principal Investigator, Emanuel João Gonçalves Ferreira de Almeida, Consultant Anesthesiologist, Hospital dos Lusíadas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CESHLAM17072023
Record Dates: First submitted 2025-12-10; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Morbid Obesity; Postoperative Pain; Opioid Free Anesthesia; Bariatric Surgery
Keywords: Opioid-free anesthesia; Bariatric surgery; Morbid obesity; Nausea and Vomiting; Postoperative pain
MeSH Terms: conditions — Obesity, Morbid; Pain, Postoperative; Nausea; Vomiting

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, two-arm parallel-group clinical trial comparing opioid-free anesthesia versus opioid-based anesthesia in patients undergoing laparoscopic bariatric surgery.
Masking Description: No blinding was implemented. Both participants and care providers were aware of group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid-Based Anesthesia (OBA) (Active Comparator): Standard opioid-based anesthesia using remifentanil infusion plus propofol induction, desflurane maintenance, and conventional multimodal analgesia, with opioids permitted for rescue.
  Interventions: Drug: Opioid-Based Anesthesia (Remifentanil-Based Protocol)
- Opioid-Free Anesthesia (OFA) (Experimental): Opioid-free anesthesia using dexmedetomidine, ketamine, and lidocaine infusion, combined with propofol induction, desflurane maintenance, and opioid-free multimodal analgesia, continued into early recovery.
  Interventions: Drug: Opioid-Free Anesthesia (Dexmedetomidine-Ketamine-Lidocaine Protocol)

INTERVENTIONS:
Drug: Opioid-Based Anesthesia (Remifentanil-Based Protocol) — Participants receive standard opioid-based general anesthesia consisting of:
  * Continuous remifentanil infusion (2 mg diluted in 40 mL saline),
  * Propofol for induction,
  * Rocuronium for neuromuscular blockade,
  * Desflurane for maintenance,
  * Dexamethasone 4-8 mg for PONV prophylaxis,
  * Cefazolin for antibiotic prophylaxis,
  * Esomeprazole for stress-ulcer prevention.
  Postoperative analgesia includes paracetamol + ketorolac/parecoxib + metamizole, with tramadol and/or morphine provided as rescue. NOL, BIS, TOF, and standard monitoring are used.
  Arms: Opioid-Based Anesthesia (OBA)
Drug: Opioid-Free Anesthesia (Dexmedetomidine-Ketamine-Lidocaine Protocol) — Participants receive opioid-free anesthesia consisting of:
  * Dexmedetomidine bolus (15-20 μg),
  * Continuous infusion of dexmedetomidine 50 μg + ketamine 50 mg + lidocaine 500 mg in 50 mL saline (rate: 1 mL/10 kg),
  * Propofol for induction,
  * Rocuronium for neuromuscular blockade,
  * Desflurane for maintenance,
  * Dexamethasone for PONV prophylaxis,
  * Cefazolin and esomeprazole for prophylaxis.
  * The analgesic infusion is reduced by half 30 min before end of surgery and continued for 1 hour in PACU.
  Postoperative analgesia includes paracetamol + ketorolac/parecoxib + metamizole, with tramadol 100 mg as rescue. Monitoring includes NOL, BIS, TOF.
  Arms: Opioid-Free Anesthesia (OFA)

SUMMARY:
This prospective randomized controlled trial aims to compare the clinical effectiveness and safety of opioid-free anesthesia (OFA) versus traditional opioid-based anesthesia (OBA) in adult patients undergoing laparoscopic bariatric surgery. The study evaluates postoperative pain, need for rescue analgesia, incidence of postoperative nausea and vomiting (PONV), intraoperative nociception monitoring (NOL index), and patient satisfaction. A total of 60 patients were randomized into two parallel groups receiving either OFA or OBA according to standardized anesthetic protocols.

DETAILED DESCRIPTION:
Bariatric surgery is the most effective treatment for severe and morbid obesity, but perioperative pain management and PONV remain significant challenges. Traditional opioid-based anesthesia is associated with adverse effects such as respiratory depression, postoperative hyperalgesia, ileus, and delayed recovery.

Opioid-free anesthesia is an emerging strategy based on the use of multimodal, non-opioid agents-including dexmedetomidine, lidocaine, and ketamine-aimed at providing adequate analgesia while reducing opioid-related complications.

This randomized controlled trial evaluates whether OFA improves postoperative pain control, reduces the requirement for rescue analgesia, and promotes better perioperative outcomes compared to OBA in laparoscopic bariatric surgery. Outcomes include NRS pain scores at multiple time points, NOL monitoring during surgery, PONV occurrence, and patient satisfaction at discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Body mass index (BMI ≥ 35 kg/m² with associated comorbidities) or BMI ≥ 40 kg/m²;
* Scheduled for elective laparoscopic bariatric surgery;
* Ability to provide informed consent.

Exclusion Criteria:

* Pregnancy;
* History of substance abuse;
* Severe psychiatric disease;
* Contraindications to any of the drugs used in either anesthetic protocol (dexmedetomidine, ketamine, lidocaine, remifentanil, etc.);
* Inability to comply with study procedures;
* Refusal or inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-21 (Actual)

PRIMARY OUTCOMES:
Postoperative pain intensity measured by the Numerical Rating Scale for Pain (NRS) | Time Frame: - Within 30 minutes of arrival at the Post-Anesthesia Care Unit (PACU); - At PACU discharge (assessed up to 2 hours after PACU admission) - Within the first 24 postoperative hours; - 48 hours postoperatively (at hospital discharge).
  Postoperative pain will be assessed using the Numerical Rating Scale for Pain (NRS), a validated 11-point scale ranging from 0 (no pain) to 10 (worst pain imaginable). Higher scores indicate a worse outcome, reflecting greater pain intensity.
  Pain intensity will be compared between the opioid-free anesthesia group and the opioid-based anesthesia group at predefined postoperative time points.

SECONDARY OUTCOMES:
Intraoperative nociception (NOL Index) | Multiple standardized time points during surgery (15 to 180 minutes)
  Nociception will be assessed using the NOL (Nociception Level) Index, a multiparametric autonomic signal-based monitor. Lower values reflect better nociceptive control. Comparisons will be made between OFA and OBA groups at all recorded time points.
Need for rescue analgesia | - During PACU stay (assessed up to 2 hours after PACU admission); - Within the first 24 postoperative hours.
  The proportion of patients requiring rescue analgesia (tramadol and/or morphine) will be compared between the opioid-free anesthesia group and the opioid-based anesthesia group.
Opioid consumption | - During PACU stay (assessed up to 2 hours after PACU admission); - Within the first 24 postoperative hours.
  Total opioid dose administered as rescue analgesia will be recorded and compared between groups.
Incidence of postoperative nausea and vomiting (PONV) | At 6 hours and 24 hours after surgery
  PONV will be assessed using the Postoperative Nausea and Vomiting Impact Scale, comparing frequency and severity between groups. The total score ranges from 0 (no nausea or vomiting) to 6 (maximum impact). Higher scores indicate a worse outcome, reflecting greater severity and clinical impact of postoperative nausea and vomiting.
Need for PONV treatment | First 24 postoperative hours
  Proportion of patients requiring antiemetic treatment will be evaluated and compared.
Patient satisfaction | 48 hours postoperatively (at hospital discharge).
  Patient satisfaction will be assessed using a Numerical Satisfaction Rating Scale and compared between groups. Total score ranges from 1 (minimum satisfaction) to 10 (maximum satisfaction). Higher scores indicate a better outcome, reflecting greater patient satisfaction.
Postoperative complications | Periprocedurally.
  Occurrence of perioperative complications (respiratory, cardiovascular, surgical, or anesthesia-related) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Emanuel J Almeida, MD, Principal Investigator — Hospital dos Lusíadas
Locations (1):
- Hospital Lusíadas Amadora - Lusíadas Saúde, S.A., Amadora, Portugal

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy restrictions and institutional regulations. Only aggregated results will be made available in publications.

DOCUMENTS (2):
  • Study Protocol (2023-07-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT07337135/Prot_000.pdf
  • Informed Consent Form (2023-07-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT07337135/ICF_001.pdf